CLINICAL TRIAL: NCT02554149
Title: Radiological Measurement of Femoral Stem Version Using Lateral Decubitus Method: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Hoi Koo, Director, Head of Orthopaedics, Principal Investigator, Professor, Seoul National University Bundang Hospital
Other Study IDs: Ante-001
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Arthroplasty; Total Hip Replacement
Keywords: total hip; stem version; replacement; hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stem anteversion: a hip lateral radiograph and CT scan were taken to measure stem anteversion
  Interventions: Radiation: Radiological measurement of femoral stem version

INTERVENTIONS:
Radiation: Radiological measurement of femoral stem version — particular radiographs( lateral decubitus view) and CT scans

SUMMARY:
The purpose of this study was to develop a radiological method to measure stem anteversion and to determine its validity and reliability.

DETAILED DESCRIPTION:
Version of the femoral stem is an important factor influencing the risk of dislocation after total hip replacement (THR) as well as the position of the acetabular component. However, there is no radiological method of measuring stem anteversion described in the literature. Investigators propose a radiological method to measure stem version and have assessed its reliability and validity. In 40 patients who underwent THR, a hip radiograph and CT scan were taken to measure stem anteversion.

ELIGIBILITY:
Inclusion Criteria:

* Investigators recruited 40 consecutive patients who underwent THR between October 2015 and December 2015

Exclusion Criteria:

* patients who could not extend the hip because of a residual flexion contracture.
* who had a flexion contracture of the knee or who could not flex the hip to 90° even after THR were excluded because participants could not adopt the posture required for the particular radiographs and CT scans.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent THR between October 2015 and December 2015
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
stem anteversion of the hip radiograph(decubitus lateral view) | postoperative 4days
stem anteversion of the CT scan | postoperative 4days

SECONDARY OUTCOMES:
The correlation between stem anteversion of the decubitus lateral view and stem version of the CT scan | postoperative 4days
  to determine ICC(intraclass coefficient, correlation coefficient)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Director, Head of Orthopaedics, Seoul National university Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeounggi-do, South Korea